CLINICAL TRIAL: NCT01512862
Title: Additive Renoprotective Effects of Oral Calcitriol in Nondiabetic Chronic Kidney Disease Patients
Brief Title: Anti-proteinuric Effect of Calcitriol in Non-diabetic Kidney Disease Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yon Su Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNUH-CCTO
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Proteinuria
Keywords: Calcitriol; Off-label
MeSH Terms: conditions — Proteinuria | interventions — Calcitriol; Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Calcitriol (Experimental)
  Interventions: Drug: Calcitriol
- Placebo (No Intervention)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcitriol — Dosage of 0.25 mcg administered orally once daily for 6 weeks and dose escalated to 0.5 mcg orally once daily up to 6 months
  Other Names: Calcio® (Hanmi Pharm Co., Korea)
  Arms: Calcitriol
Drug: Placebo — Dosage of 0.25 mcg administered orally once daily for 6 weeks and dose escalated to 0.5 mcg orally once daily up to 6 months
  Arms: Placebo

SUMMARY:
Proteinuria is not only a marker of chronic kidney disease (CKD) progression, but also a marker of cardiovascular disease and death. In previous studies, active vitamin D deficiency is associated with cardiovascular risk factors such as albuminuria, diabetes mellitus, and lower glomerular filtration rate (GFR). And calcitriol was shown to have a preventive effect in progressive glomerular damage in a renal ablation model. Calcitriol, an active form of vitamin D (1,25-dihydroxyvitamin-D3), is commonly used for the treatment of secondary hyperparathyroidism in patients with advanced chronic kidney diseases.

Therefore, the objective of this study is to evaluate the anti-proteinuric effect of calcitriol in non-diabetic kidney disease patients. They will be treated with calcitriol and placebo for 24 weeks and observed for 24 weeks after treatment. Proteinuria, renal function, serum and urinary inflammatory markers, and adverse event will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Nondiabetic kidney disease patients aged 19-70 years
* MDRD GFR ≥ 30 mL/min/1.73m2
* Patients with residual urine protein/creatinine ratio > 200 mg/g
* Adequate blood pressure control as treated systolic blood pressure <=140 or diastolic <=90 mmHg with RAS inhibitor for more than 3 months
* Normotensive patients untreated with RAS inhibitors
* Serum intact PTH as 35-500 mg/dL and serum calcium less than 10.2 mg/dL
* Patients who have not been treated vitamin D within the 3 months prior to signing the informed consent form

Exclusion Criteria:

* Patients with nephrotic-range proteinuria (24 hour urine protein >3.5 g/24 hr)
* Patients with rapidly progressive glomerulonephritis
* Patients requiring renal replacement therapy immediately
* Hypercalcemia (uncorrected serum calcium level > 10.2 mg/dL) within 3 months
* Malignant hypertension
* Heart failure (New York Heart Association [NYHA] functional class II to IV or LVEF less than 40%)
* Severe chronic obstructive lung disease
* Decompensated liver disease
* Known allergy or hypersensitivity to vitamin D
* Current treatment with steroids and/or immunosuppressive agents
* No other active primary malignancy requiring treatment or that limits survival to ≤ 2 years
* History of noncompliance to medical regimen
* Inability to give an informed consent or to cooperate with researchers (e.g., psychiatric disorder)

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Changes in proteinuria | 6, 12 months after administration
  Comparison of proteinuria amount checked by random urine protein/creatinine ratio

SECONDARY OUTCOMES:
Changes in renal function | 3, 6, 9 and 12 months
  Comparison of in serum creatinine level from baseline
Changes in urinary renal damage markers | 6, 12 months
  Comparison of urinary TGF-beta, TNF-alpha, MCP-1 level from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jung Mi Oh, Pharm.D., Study Chair — Seoul National Univerisy College of Pharmacy; Yon Su Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul